CLINICAL TRIAL: NCT01321814
Title: Cognitive Behavioral Therapy for Hyperacusis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Uppsala University (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GA-LJ-HYP1
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Hyperacusis
Keywords: Hyperacusis; Personality; Comorbidity; Treatment; Cognitive behavioral therapy
MeSH Terms: conditions — Hyperacusis | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioural therapy (CBT) (Experimental): Patients receiving 6 sessions of CBT conducted by a licensed psychologist. Sessions include psychoeducation, exposure treatment, behavioral activation and applied relaxation.
  Interventions: Behavioral: Cognitive behavioural therapy
- Waiting list (No Intervention): Patient waits for CBT treatment for 6 months.

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy — 6 sessions by licensed psychologist, including psychoeducation, exposure therapy, applied relaxation and behavioral activation.
  Arms: Cognitive behavioural therapy (CBT)

SUMMARY:
The main purpose of this study is to investigate whether cognitive behaviour therapy (CBT) can be useful for people suffering from Hyperacusis.

Also, the investigators are interested in investigating this group of patients on psychiatric and somatic comorbidity, personality traits, and startle response to sounds.

The investigators will also study the audiological measures commonly used in Sweden to measure hyperacusis, and investigate their validity.

The investigators hypothesize that CBT might be helpful for patients suffering from Hyperacusis.

DETAILED DESCRIPTION:
Hyperacusis, defined as unusual intolerance to ordinary environmental sounds, is a common problem for which there are no controlled trials on psychological treatment. Given the avoidance strategies present in hyperacusis, and similarities with problems such as tinnitus and chronic pain, cognitive behaviour therapy (CBT) is hypothesized to be helpful for patients with hyperacusis. In this randomized controlled study of 60 patients with hyperacusis, CBT was compared with a waiting list control group using the Loudness Discomfort Level test (LDL), the Hyperacusis Questionnaire, the Hospital Anxiety and Depression Scales, the Quality of Life Inventory and an adapted version of the Tampa Scale of Kinesiophobia. There were significant between-group effects in favour of the CBT group on all measures except for the HADS anxiety scale. Between-group effect sizes were moderate to high, with Cohen's d = 0.67 and 0.69 per ear, respectively, for the primary measure LDL, and ranging from d = 0.32 to 1.36 for the secondary measures. The differences between groups ceased to exist when the waiting list group was treated later with CBT, and the treatment results were largely maintained after 12 months. In conclusion, CBT is a promising treatment for hyperacusis, although more research is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patient understands and can speak Swedish well
* Hyperacusis is the primary audiological problem
* Loudness discomfort thresholds below 90 dB
* Hearing levels better than 40dB on the best ear
* Resident of Uppsala, Stockholm or Vastmanland
* Possibility to travel to Uppsala or Vasteras for examination and treatment

Exclusion Criteria:

* Scoring "moderate" or "high" on suicidality, according to M.I.N.I
* Moderate to severe depression
* Psychotic disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-06; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life Inventory (QOLI) | Evaluation for participance (day one), before treatment for waiting list patients (up to 6 months), direct after treatment, 12 mts after treatment
  Inventory measuring how patients' percieve the importance of and their satisfaction with many variables that concludes life quality, for instance economy, physical health and family life.
Khalfa Hyperacusis Questionnaire | Evaluation for participance (day one), before treatment for waiting list patients (up to 6 months), direct after treatment, 12 mts after treatment
  A questionnaire to quantify and evaluate various hyperacusis symptoms, screening several aspects of auditory symptomatology.
Loudness discomfort threshold | Time Frame: (FDAAA) Evaluation for participance (day one), before treatment for waiting list patients (up to 6 months), direct after treatment, 12 mts after treatment
  Audiological measure where the patient is exposed to sounds, gradually of higher volume. The patient is instructed to indicate when the sound level is uncomfortably loud, and that terminates the exposure. The test is performed by an audiologist using a calibrated audiometer.

SECONDARY OUTCOMES:
The Mini-International Neuropsychiatric Interview (M.I.N.I) | At evaluation for participance (day one)
  M.I.N.I is a short structured diagnostic interview (Sheehan et al, 1998), developed to detect DSM-IV and ICD-10 psychiatric disorders and was performed to investigate psychiatric comorbidity in this study. The Swedish version, 5.0.0. was used.
Swedish universities Scales of Personality (SSP) | At evaluation for participance (day one)
  SSP aims to measure personality correlates as well as biological correlates of some psychiatric disorders in order to define vulnerability factors (Gustavsson et al, 2000). The test consists of 13 scales, for instance somatic trait anxiety, psychic trait anxiety and stress susceptibility.
Tampa scale of Kinesiophobia - for Hyperacusis | Evaluation for participance (day one), before treatment for waiting list patients (up to 6 months), direct after treatment, 12 mts after treatment
  TSK is a questionnaire used to measure fear of movement or reinjury in chronic pain patients. For this study, we adapted TSK for Hyperacusis patients.
Startle-response | Evaluation for participance (day one), before treatment for waiting list patients (up to
  Heart rate and skin conductance measured in response to sounds, in level with LDL:s.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ekselius, Professor, Study Director — Uppsala University; Gerhard Andersson, Professor, Study Chair — Linkoeping University; Hans C Larsen, Reader, Study Chair — Uppsala University Hospital; Linda Jüris, PhD Student, Principal Investigator — Uppsala University/ Uppsala University Hospital
Locations (1):
- Uppsala, Sweden